CLINICAL TRIAL: NCT04901767
Title: Comparison of Intracoronary Endothelial Dysfunction in Patients With Coronary Artery Disease Treated With Drug Coated Balloon Angioplasty and Drug Eluting Stents
Brief Title: Coronary Artery Endothelial Dysfunction With Drug Coated Balloons
Acronym: SPARTAN-VM
Status: Completed | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 262024 (207-11-19)
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Ischaemic Heart Disease; Endothelial Dysfunction
Keywords: Percutaneous coronary intervention; Drug coated balloons; Drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Receiving drug coated balloon (DCB)
- Receiving drug eluting stent (DES)

SUMMARY:
Use of intracoronary acetylcholine to investigate endothelial function in coronary arteries treated with either drug coated balloon angioplasty of drug eluting stents.

DETAILED DESCRIPTION:
The primary objective is to establish the differences in vasomotor response of a DCB and DES treated artery by measurement of the percentage change in coronary surface area pre and post acetylcholine administration. This will be measured with incremental doses of acetylcholine at levels both proximally and distally to the site of treatment Also is to see how far endothelial dysfunction may propagate from an interventional site by measuring drug induced dilatation/constriction as in response to acetylcholine administration. This vasomotor response will be measured in the target vessel at extended distances from the treated segment.

To achieve a meaningful comparison, 34 patients will be recruited of which 17 patients would form either arm of the study having had either a DCB or DES.

The study will be performed at the Norfolk and Norwich University Hospital and patients will be enrolled prior to a second procedure. This may occur immediately after their stent or drug coated balloon treatment or if they re-attend hospital in the following recruitment period and this may include patients for a variety of different indications.

Patients who have a scheduled, clinically indicated procedure will be eligible to be recruited as participants. They must also fulfil the inclusion criteria and not be affected by any of the exclusion criteria.

A member of the research team will provide the Patient Information Sheet to potential participants and confirm that they would be happy to be contacted subsequently to discuss the proposed research. The subsequent contact will be undertaken by a clinical research fellow, who is both a member of the Norfolk and Norwich University Hospital NHS clinical team as well as the research team, prior to their subsequent visit to discuss the study, answer any questions and confirm if they fulfil the inclusion criteria. In view of Covid-19, to reduce in hospital exposure, we might instead opt to send the patient information to the eligible patients by post, and follow with a telephone call to confirm receipt.

Method: Patients will be prepared in the usual way as per clinical practice for their procedure. They will attend via a standardised case pathway depending on the indication for repeat angiography (staged procedure versus re-presentation acutely for another reason such as chest discomfort). There are a series of routine checks performed to ensure that the patient is on appropriate medications. For the purpose of the study, anti-anginal medications will need to be stopped for 72 hours prior to the procedure. The anti-anginal medications that would require cessation include:

* Cardio selective Beta 1 selective blockers (Atenolol, Bisoprolol, Carvedilol, Esmolol, Metoprolol and Nebivolol )
* Diltiazem
* Nicorandil
* Isosorbide Nitrate preparations
* Ranolazine The particular medication regime will vary on a patient to patient basis and the appropriateness of this and nature of drug cessation will be discussed at the enrolment process and patients will be given clear instruction on adjustments to their regimen.

Coronary Angiography will be performed as per common clinical practice. At the beginning of the study portion of the procedure, there will be two orthogonal angiographic views taken of the treated segment which will then be denoted as the reference views for the rest of the procedure (used after every administration of agonist).

Acetylcholine (ACh) will be diluted into 0.9% normal saline at different dilutions (to a total volume of 5mL). NB - these solutions of Acetylcholine are usable within a two-hour period, beyond this time a new solution should be used. When reassessing the previously treated artery, an infusion of intracoronary acetylcholine will be administered via the guiding catheter. The first ACH infusion ("low dose") will be 0.182micrograms/mL (10^-6mol/L) given at a rate of 1Ml/min for two minutes by a mechanical infusion pump (50). After the infusion, intracoronary contrast will be injected and images acquired.

If there are no adverse features, the investigator can proceed with the subsequent increments with each infusion to complete, followed by a five-minute interval. The next increments would be:

* "medium dose" 1.82mcg/ml (10^-5mol/L) ACH in 5ml normal saline - given over 20 seconds.
* "high dose" 18.2mcg/ml (10^-4mol/l) ACH in 5ml normal saline - given over 20 seconds.
* Then after a further five minutes - a bolus dose of GTN (400mcg) will be administered over 20 seconds and then a further contrast acquisition taken within two minutes. Also see Appendix C for lab flow chart.

Once these images have been taken, the guide catheter will be removed the procedure will then be completed in the usual way. The patient with then be moved to the appropriate recovery area as per the standard protocol following PCI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Been treated with percutaneous coronary intervention of either drug coated balloon or drug eluting stent

Exclusion Criteria:

* Any contraindications to administration of acetylcholine or GTN
* History of coronary vasospasm or spontaneous coronary artery dissection
* Significant medical, surgical or psychiatric disease that would affect subject safety or influence the study outcome according to physician's opinion
* Patients who received a combination of drug eluting stents and drug coated balloon to the same vessel
* Significant renal impairment (estimated glomerular filtration rate <30mL/min/ 1.73m2
* Body mass index >35 (may affect coronary artery diameter qualitative assessment)
* Symptomatic congestive cardiac failure
* Severe asthma
* Significant autoimmune inflammatory conditions (for example rheumatoid arthritis)
* Patients taking immunomodulating drugs (including Methotrexate, Ciclosporin, steroids)
* Previous heart transplant
* Relative Anaemia - Haemoglobin <12g/dL in men and <10g/dL in women
* Women of child bearing age with a positive pregnancy test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be included who have received percutaneous coronary intervention with either a drug coated balloon or drug eluting stent and stable symptoms. Patients who have a clinically indicated procedure will be eligible to be recruited as participants. They must also fulfil the inclusion criteria and not be affected by any of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Fractional change in coronary artery diameter and surface area within treated segment | 3-6 months
  Will be expressed as a percentage. I.e. we will measure the diameter in mm and area in mm2 before and after.

SECONDARY OUTCOMES:
Fractional change in coronary artery diameter and surface area with increments from area of treatment | 3-6 months
  Will be expressed as % rather than units.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Dr Merinopoulos, Study Chair — IOANNIS.MERINOPOULOS@nnuh.nhs.uk; Vassilis Dr Vassiliou, Principal Investigator — VASSILIOS.VASSILIOU@nnuh.nhs.uk
Locations (1):
- Norfolk & Norwich University Hospital, Norwich, Norfolk, United Kingdom

REFERENCES:
- See also: Dysfunction</b> Int Heart J [Internet]. 2007;48(5):553-67. — http://www.jstage.jst.go.jp/article/ihj/48/5/48_5_553/_article
- See also: Koskinas KC, Chatzizisis YS, Antoniadis AP, Giannoglou GD. Role of Endothelial Shear Stress in Stent Restenosis and Thrombosis. J Am Coll Cardiol [Internet]. 2012;59(15):1337-49. — http://dx.doi.org/10.1016/j.jacc.2011.10.903
- See also: Ohtsuka M, Yokoyama S, Imaizumi T, Mitsutake Y, Toyama Y, Chibana H, et al. Coronary Endothelial Dysfunction Distal to Stent of First-Generation Drug-Eluting Stents. JACC Cardiovasc Interv [Internet]. 2012;5(9):966-73. — http://dx.doi.org/10.1016/j.jcin.2012.06.010
- See also: Ho HH, Ong PJL. BASKET-SMALL 2: advancing DCB beyond in-stent restenosis. Lancet [Internet]. 2018;392(10150):802-4. — http://dx.doi.org/10.1016/S0140-6736(18)31926-3